CLINICAL TRIAL: NCT05520502
Title: The Effect of Pilates exercıses on Engine Performance and Body Composition ın Primary School Children
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Suleyman Demirel University (Other)
Responsible Party: Principal Investigator, Handan Çağlar Çavdar, lecturer, Suleyman Demirel University
Other Study IDs: 72867572
Record Dates: First submitted 2022-07-21; First posted 2022-08-30 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Exercise; Body Weight Changes
Keywords: EXERCISE; PERFORMANCE; PILATES EXERCISE; BODY COMPOSİTİON; CHILDREN
MeSH Terms: conditions — Motor Activity; Body Weight Changes | interventions — Exercise Movement Techniques

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: PILATES EXERCISE — 12 WEEKS, 3 SESSIONS A WEEK 36 SESSIONS IN A TOTAL OF PLANNED MAT 1 PILATES EXERCISES

SUMMARY:
In thıs study, planned for prımary chıldren between 7-11 years, pılates exercıses wıll be done wıth the chıldren who accept to partıcıpate ın the study wıth the accountance of the researcher and compared wıth the control group. Evaluatıon; parameters; engıne performance tests and body composıtıon analysıs.

DETAILED DESCRIPTION:
It is a fact that there are disadvantages as well as advantages brought by the development of technology. With this development, individuals adopt a more sedentary lifestyle and daily physical activity and mobility are gradually decreasing. These deficiencies have affected the child population as much as adults. This lack of physical activity in childhood negatively affects the child's growth, development, mood and school success, and increases the risk of chronic diseases in adulthood by preparing the ground for obesity.

The positive effects of physical activity on human health are multifaceted. Physical, mental, social and cognitive well-being is among its well-known benefits. Especially the physical activity and exercise habits gained in childhood contribute greatly to the mental, physical and emotional development of children.

The positive effects of the Pilates method on individuals' muscular strength and endurance, motor performance and body composition have been reported in many studies. Pilates exercise method is a suitable and reliable type of physical activity that can be done for children, and it has positive contributions to the growth, development and postural development of children .

Our aim in this study, which we will do with 7-11 age group primary school children, is to investigate the effects of regular physical activity and exercise, such as pilates, on both motor ability and body composition.

Our hypotheses in our study;

H1: Pilates exercises improve motor ability in primary school children. H2: Pilates exercises positively affect body composition in primary school children H3: Pilates exercises do not affect motor ability in primary school children. H4: Pilates exercises do not affect body composition in primary school children.

Pilates studies with healthy children are not common in our country. Therefore, our study is the first long-term planned (12 weeks 36 sessions) pilates study to be carried out with healthy children at primary school age.

Apart from this, when looking at the evaluation parameters, criteria such as pain, physical fitness, balance were frequently investigated with pilates.

Apart from these, motor ability tests and body composition analysis with a bioimpedance body analyzer will be evaluated in our study, and in this sense, it is one of the first pilates studies conducted with healthy children with these parameters.

ELIGIBILITY:
Inclusion Criteria:

* AGREEING TO PARTICIPATE IN THE STUDY,
* NO CHRONIC DISEASE,
* NO SPORTS HISTORY

Exclusion Criteria:

* Failing to COMPLETE SESSIONS
* PRESENCE OF CHRONIC DISEASE
* Engaging in SPORTS ACTIVITIES

Ages: 7 Years to 11 Years | Sex: All
Age Groups: Child
Study Population: primary school chilrens
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2022-02-14 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
The effect of pilates exercıses on engine performance and body composition ın primary school children | february 2022- september 2022
  STUDY GROUP EXERCISE PERIOD IS NOT OVER
BODY MASS INDEX | february 2022- september 2022
  KG/M2

OTHER OUTCOMES:
PERFORMANCE TESTS | february 2022- september 2022

CONTACTS AND LOCATIONS:
Locations (1):
- Süleyman Demirel Üniversitesi, Isparta, Turkey (Türkiye)